CLINICAL TRIAL: NCT01658475
Title: Assessment of Use of Plasma or Serum IgG Test to Screen for Periodontitis
Brief Title: P. Gingivalis IgG Titer Test for Periodontitis
Status: Completed | Type: Observational
Sponsor: Okayama University (Other)
Responsible Party: Principal Investigator, Shogo Takashiba, Professor and Chair, Okayama University
Other Study IDs: OUGSMDPS-350&453; JSPS #18209061 & H19-Choju-008 (Other Grant/Funding Number: JSPS & Ministry of Health, Labor, and Welfare of Japan)
Record Dates: First submitted 2012-07-31; First posted 2012-08-07 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Periodontitis
Keywords: IgG titer; periodontopathic bacteria
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma and/or serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- periodontitis: those with periodontitis and those without periodontitis

SUMMARY:
This study was performed to evaluate prospectively the diagnostic utility of a blood IgG antibody titer test against periodontal pathogens.

DETAILED DESCRIPTION:
Background: Periodontitis is a prevalent silent infectious disease worldwide, and affects lifestyle-related diseases such as diabetes. Therefore, efficient screening of patients is essential for general health. This study was performed to evaluate prospectively the diagnostic utility of a blood IgG antibody titer test against periodontal pathogens.

Methods: Oral examination was performed and blood IgG antibody titers against periodontal pathogens were measured by ELISA, in 1387 subjects. The cut-off value of IgG titer was determined in receiver operating characteristic curve analysis, and changes in periodontal clinical parameters and IgG titers by periodontal treatment were evaluated. The relationships between IgG titers and severity of periodontitis were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* periodontal patients
* adults

Exclusion Criteria:

* difficulty of communication
* received periodontal therapy within 3 months
* with other diseases, i.e., hypertension, diabetes (self reported)

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who visit university hospitals to receive periodontal treatment are patients group.
  Employees who receive occupational health check at a company facility.
Sampling Method: Non-Probability Sample
Enrollment: 1387 (Actual)
Dates: Start 2007-01; Primary Completion 2009-11 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Level of IgG antibodies in serum/plasma against periodontal pathogens | 1 to 3 months after basic periodontal treatment (Scaling and root planing)
  Serum/plasma samples will be screened for the presence of IgG antibodies against the below mentioned periodontal pathogens, using the "ELISA" method.
  Aggregatibacter actinomycetemcomitans, Eikenella corrodens, Prevotella intermedius, Porphyromonas gingivalis

SECONDARY OUTCOMES:
Periodontal pocket depth | 1 to 3 months after basic periodontal treatment
  Clinical observation on periodontal pocket depth before and after basic periodontal treatment, in order to confirm appropriate effects of the treatment.
Bleeding on probing | 1 to 3 monthsafter basic periodontal treatment
  Judging from bleeding from gingiva after periodontal pocket probing, degree of inflammation will be understood.
Tooth mobility | 1 to 3 months after basic periodontal treatment
  Clinical observation to understand decrease of inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Shogo Takashiba, Professor, Principal Investigator — Okayama University Graduate School of Medicine, Dentistry and Pharmaceutical Sciences, Department of Pathiphysiology - Periodontal Science
Locations (12):
- Japan (12):
  - Aichi Gakuin University, School of Dentistry, Nagoya, Aichi-ken
  - Toyota Motor Corporation, Toyota, Aichi-ken
  - Nihon University School of Dentistry at Matsudo, Matsudo, Chiba
  - Hiroshima University Graduate School of Biomedical Sciences, Hiroshima, Hiroshima
  - Tohoku University Graduate School of Dentistry, Sendai, Miyagi
  - Nagasaki University Graduate School of Biomedical Sciences, Nagasaki, Nagasaki
  - Niigata University Faculty of Dentistry, Niigata, Niigata
  - Okayama University Graduate School of Medicine, Dentistry and Pharmaceutical Sciences, Okayama, Okayama-ken
  - Osaka University Graduate School of Dentistry, Suita, Osaka
  - The University of Tokushima Graduate School, Institute of Health Biosciences, Tokushima, Tokushima
  - Tokyo Medical and Dental University Graduate School, Bunkyo-ku, Tokyo
  - Nippon Dental University, School of Life Dentistry at Tokyo, Chiyoda-ku, Tokyo

REFERENCES:
- [Derived] Kudo C, Naruishi K, Maeda H, Abiko Y, Hino T, Iwata M, Mitsuhashi C, Murakami S, Nagasawa T, Nagata T, Yoneda S, Nomura Y, Noguchi T, Numabe Y, Ogata Y, Sato T, Shimauchi H, Yamazaki K, Yoshimura A, Takashiba S. Assessment of the plasma/serum IgG test to screen for periodontitis. J Dent Res. 2012 Dec;91(12):1190-5. doi: 10.1177/0022034512461796. Epub 2012 Sep 26. PMID 23018816
- See also: Introduction site for the project supported by JSPS, and guiding the visitors to "Web-based Management System for Data of Periodontal Infection". Notice: this site is written in Japanese. — http://www.cc.okayama-u.ac.jp/~perio/stakashi_web/kiban_a_site/index.html